CLINICAL TRIAL: NCT02617511
Title: Omega-3 Fatty Acid Supplementation and Resistance Training on Inflammation and Body Composition in Older Men
Brief Title: Omega-3 Supplementation and Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2015:020
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2015-11

CONDITIONS: Sarcopenia; Dynapenia; Inflammation
MeSH Terms: conditions — Sarcopenia; Inflammation | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids; Linseed Oil; Rapeseed Oil; black currant oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Supplementation (Experimental): This groups will supplement their regular diet with 2.97 grams of combined omega-3 fatty acid (EPA/DHA) supplement in soft gel form on a daily basis for 12 weeks. This group will also complete a whole body progressive resistance training program 3 days per week for 12 weeks.
  Interventions: Dietary Supplement: Omega-3 Supplementation
- Placebo (Placebo Comparator): This group will supplement their regular diet with 3.0 grams of a combined omega-3-6-9 supplement in soft gel form on a daily basis for 12 weeks. This group will also complete a whole body progressive resistance training program 3 days per week for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Supplementation
  Other Names: eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)
  Arms: Omega-3 Supplementation
Dietary Supplement: Placebo
  Other Names: flax seed oil, evening primrose oile, canola oil, black currant oil, pumpkin seed oil
  Arms: Placebo

SUMMARY:
The purpose of this project is to evaluate whether omega-3 fatty acid supplementation (combined eicosapentaenoic acid and docosahexaenoic acid [EPA/DHA] supplement) augments the effects of a 12-week resistance training program in older men. Outcome variables include inflammatory biomarkers in the systemic circulation, body composition and performance measures. The specific inflammatory markers in the blood include: C-reactive protein, tumor necrosis factor-α, interleukin-1β, and interleukin-6. Remaining parameters include: body composition (as assessed by dual energy x-ray absorptiometry), muscle strength (as assessed by chest press and leg press one-repetition maximum strength tests), and functional ability (as assessed by timed up and go test as well as the 6-minute walking test).

DETAILED DESCRIPTION:
Summary: Sarcopenia is a prevalent health concern for many older individuals and finding strategies to ameliorate and reduce the loss of skeletal muscle mass and strength is deemed important for maintaining functional ability and independence as individual's age. Currently, resistance training is considered the standard of care for inducing an anabolic stimulus and preserving as well as enhancing muscle mass and strength in aged individuals. One mechanism whereby older adults seem to lose muscle mass with age is via chronic low grade inflammation. Finding complementary strategies to reduce inflammation, while at the same time building skeletal muscle mass and strength, is considered essential for combating the increased prevalence of sarcopenia observed as the population ages. Using nutritional supplementation strategies, such as omega-3 fatty acids, seems to provide an effect in not only reducing inflammation but also acting as an anabolic stimulus for skeletal muscle growth. It is not known whether or not providing omega-3 fatty acids (in the form of EPA/DHA supplementation) along with resistance training will result in a greater increase in skeletal muscle mass and strength than resistance training alone in an older population.

Hypotheses: The primary hypothesis of this research project is that omega-3 fatty acid supplementation and resistance training for 12 weeks will decrease markers of inflammation more so than resistance training and placebo in a cohort of older adults. A secondary hypothesis of the project is that omega-3 fatty acid supplementation and resistance training for 12 weeks will provide for a greater increase in skeletal muscle mass, strength, and functional ability than resistance training and placebo in a cohort of older adults.

ELIGIBILITY:
Inclusion Criteria:

1. equal to or greater than 65 years of age,
2. male,
3. they will not participate in a structured exercise program any more than 2-times per week.

Exclusion Criteria:

1. consumption of anti-inflammatory medication (which would confound the results in terms of the effects that the exercise and nutritional intervention is accomplishing),
2. diagnosis with an inflammatory disease (such as inflammatory bowel disease or rheumatoid arthritis) as this is not the participant population we want to evaluate,
3. consumption of any natural health products that have anti-inflammatory components to them (such as omega-3 fatty acids or omega-3 fortified eggs or more than 2 servings per week of fatty fish),
4. current participation in an exercise program ≥ 2 times per week or current participation in a structured resistance training program > 1 time per week as we want to evaluate an untrained, sedentary population,
5. has a mental or cognitive disability (such as dementia), and
6. has a physical disability that would limit them from participating in a structured resistance training program.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Cornish, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- Applied Research Centre, Faculty of Kinesiology, University of Manitoba, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Omega-3 Supplementation: This groups will supplement their regular diet with 2.97 grams of combined omega-3 fatty acid (EPA/DHA) supplement in soft gel form on a daily basis for 12 weeks. This group will also complete a whole body progressive resistance training program 3 days per week for 12 weeks.
  Omega-3 Supplementation
- Placebo: This group will supplement their regular diet with 3.0 grams of a combined omega-3-6-9 supplement in soft gel form on a daily basis for 12 weeks. This group will also complete a whole body progressive resistance training program 3 days per week for 12 weeks.
  Placebo
Period: Overall Study
Arm/Group | Omega-3 Supplementation | Placebo
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Older males (>/= 65 years of age)
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Supplementation | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (6.2) | 70.9 (5.0) | 71.1 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 12 | 23
Baseline Characteristics [Mean (Standard Deviation); unit: Height (cm)] | 175.1 (4.7) | 176.7 (5.7) | 175.9 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Necrosis Factor-alpha
Description: The cytokine tumor necrosis factor-alpha will be used as the primary outcome to assess change in inflammatory status over the 12 week intervention
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Omega-3 Supplementation | Placebo
Number analyzed (Participants) | 11 | 12
pg/mL
  Baseline | 1.05 (0.49) | 0.93 (0.54)
  12 weeks post | 1.04 (0.41) | 1.18 (0.59)

2. Secondary Outcome: Interleukin-6
Description: Interleukin-6 will be used to assess changes in inflammatory status.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Omega-3 Supplementation | Placebo
Number analyzed (Participants) | 11 | 12
pg/mL
  Baseline | 2.01 (1.49) | 1.84 (0.93)
  12 weeks post | 2.1 (1.49) | 2.19 (1.21)

3. Secondary Outcome: Lean Tissue Mass
Description: Dual energy x-ray absorptiometry will be used to assess changes in lean tissue mass.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Omega-3 Supplementation | Placebo
Number analyzed (Participants) | 11 | 12
kilograms
  Baseline | 55.2 (6.3) | 55.8 (6.1)
  12 weeks post | 55.7 (5.9) | 56.5 (5.6)

4. Secondary Outcome: Leg Press Strength
Description: A one-repetition maximum leg press strength test will be used to assess lower body strength.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Omega-3 Supplementation | Placebo
Number analyzed (Participants) | 11 | 12
kilograms
  Baseline | 114.5 (38.4) | 105.7 (27.8)
  12 weeks post | 158.7 (50) | 142.0 (31.2)

5. Secondary Outcome: Timed up and go Test
Description: Mobility and balance will be assessed using a 3 meter timed up and go test.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Omega-3 Supplementation | Placebo
Number analyzed (Participants) | 11 | 12
seconds
  Baseline | 6.35 (1.06) | 5.91 (0.58)
  12 weeks post | 5.83 (1.11) | 5.62 (0.44)

6. Secondary Outcome: Bone Mineral Content
Description: Dual energy x-ray absorptiometry will be used to assess changes in bone mass.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Omega-3 Supplementation | Placebo
Number analyzed (Participants) | 11 | 12
kilograms
  Baseline | 3.18 (0.31) | 3.26 (0.15)
  12 week post | 3.19 (0.31) | 3.26 (0.16)

7. Secondary Outcome: Chest Press Strength
Description: A one-repetition maximum chest press strength test will be used to assess upper body strength.
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Omega-3 Supplementation | Placebo
Number analyzed (Participants) | 11 | 12
kilograms
  Baseline | 51.4 (19.6) | 49.6 (14.3)
  12 weeks post | 67.2 (25.1) | 65.0 (13.9)

8. Secondary Outcome: 6 Minute Walk Test
Description: A 6 minute walk test will be used to assess the distance walked in 6 minutes of continuous walking.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Omega-3 Supplementation | Placebo
Number analyzed (Participants) | 11 | 12
meters
  Baseline | 604.8 (71.1) | 622.5 (43.6)
  12 weeks post | 636.7 (89.8) | 646.4 (64.6)

ADVERSE EVENTS:
Arm/Group | Omega-3 Supplementation | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Supplementation (N=11) | Placebo (N=12)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No